CLINICAL TRIAL: NCT03304522
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, 6-Week, Parallel-design Study of the Efficacy and Safety of VX-150 in Treating Subjects With Pain Caused by Small Fiber Neuropathy
Brief Title: A Study to Evaluate the Efficacy and Safety of VX-150 in Treating Subjects With Pain Caused by Small Fiber Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX16-150-102; 2017-001042-10 (EudraCT Number)
Record Dates: First submitted 2017-09-18; First posted 2017-10-09 (Actual); Results first posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Small Fiber Neuropathy
MeSH Terms: conditions — Small Fiber Neuropathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VX-150 (Experimental)
  Interventions: Drug: VX-150
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VX-150 — Participants received VX-150 1250 milligrams (mg) once daily (qd) orally for 6 weeks.
  Arms: VX-150
Drug: Placebo — Participants received placebo matched to VX-150 for 6 weeks.
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled, parallel-group, multicenter study evaluating the efficacy of VX-150 for the treatment of pain caused by small fiber neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 31.0 kg/m2, inclusive, and a total body weight >50 kg
* Diagnosis of small fiber neuropathy, as per European Federation Neurological Societies (EFNS)/American Academy of Neurology (AAN) guidelines, with pain for at least 3 months prior to screening
* Reduction below the 5th percentile of sex and age-adjusted normal values in epidermal nerve fiber density on punch skin biopsy at the distal site of the leg performed at screening
* Normal nerve conduction studies (NCS), including presence of sural response.
* Average NRS score between ≥4 and ≤9 reported in the daily diary on Days -7 through -1

Exclusion Criteria:

* History in the past 10 years of malignancy except for squamous cell skin cancer, basal cell skin cancer, and Stage 0 cervical carcinoma in situ
* History of connective tissue disorders, sarcoidosis, Sjögren's syndrome, amyloidosis, Fabry's disease, celiac disease, lyme disease, autoimmune disorders
* A known or clinically suspected infection with human immunodeficiency virus or hepatitis B or C viruses
* Current clinically significant liver or kidney dysfunction
* Current uncontrolled thyroid dysfunction
* A diagnosis of diabetes, HbA1C ≥8% at screening
* History of cardiac dysrhythmias requiring anti-arrhythmia treatment(s)
* Concomitant severe pain conditions which may impair self-assessment of pain due to small fiber neuropathy

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2018-11-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (31):
  - Xenoscience Inc. - 21st Century Neurology, Phoenix, Arizona
  - Phoenix Neurological Associates, Ltd., Phoenix, Arizona
  - Sutter Health - Alta Bates Summit Medical Center - The Jordan Research & Education Institute, Berkeley, California
  - Neuropain Medical Center, Fresno, California
  - University of California San Diego, La Jolla, California
  - SDS Clinical Trials, Inc., Orange, California
  - Stanford University School of Medicine, Redwood City, California
  - Blue Sky Neurology, Englewood, Colorado
  - Bioclinica Research - Orlando, Orlando, Florida
  - Infinity Clinical Research, Sunrise, Florida
  - Southern Illinois University (SIU) School of Medicine, Springfield, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center (KUMC), Kansas City, Kansas
  - International Clinical Research Institute (ICRI), Overland Park, Kansas
  - River Cities Clinical Research Center, Shreveport, Louisiana
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center (DHMC), Lebanon, New Hampshire
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - Albany Medical Center- Neurology Group, Albany, New York
  - The Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Duke Neurological Disorders Clinic, Durham, North Carolina
  - Carolinas Pain Institute, Winston-Salem, North Carolina
  - Neurology Diagnostics, Inc, Dayton, Ohio
  - The Richter Clinic for Neurology and Neuro-Psychiatry, Tulsa, Oklahoma
  - Carilion Clinic Neurology, Roanoke, Virginia
  - University of Washington, Seattle, Washington
- Universitätsklinikum Würzburg, Würzburg, Germany
- Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta, Milan, Italy
- Maastricht UMC+, Maastricht, Netherlands

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 89 participants were enrolled and randomized in the study.
Groups:
- VX-150: Participants received VX-150 1250 milligram (mg) once daily (qd) for 6 weeks.
Period: Overall Study
Arm/Group | VX-150 | Placebo
Started | 46 | 43
Completed | 45 | 35
Not Completed | 1 | 8
Not completed — Adverse Event | 0 | 4
Not completed — Withdrawal of consent (due to lack of efficacy) | 1 | 1
Not completed — Withdrawal of consent (for other reason) | 0 | 2
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- VX-150: Participants received VX-150 1250 mg qd for 6 weeks.
- Total: Total of all reporting groups
Arm/Group | VX-150 | Placebo | Total
Number analyzed (Participants) | 46 | 43 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (12.34) | 58.1 (11.86) | 56.6 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 24 | 22 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 43 | 38 | 81
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 39 | 34 | 73
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 2 | 2
Pain Intensity at Baseline on 11-point Numeric Rating Scale (NRS) [Mean (Standard Deviation); unit: units on a scale] — Pain intensity was evaluated using the 11-point NRS (where 0 signified no pain and 10 signified worst imaginable pain). Higher score indicates greater level of pain. Baseline score was average of daily pain scores from Day -7 to Day -1.
  units on a scale | 6.433 (1.440) | 5.990 (1.413) | 6.219 (1.436)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weekly Average of Daily Pain Intensity on the 11 Point NRS
Description: Pain intensity was evaluated using the 11-point NRS (where 0 signified no pain and 10 signified worst imaginable pain) during the last 24 hours on the NRS each evening. Higher score indicates greater level of pain.
Time Frame: From Baseline at Week 6
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | VX-150 | Placebo
Number analyzed (Participants) | 46 | 43
units on a scale | -2.018 (0.274) | -0.933 (0.287)
Statistical Analysis 1: Comparison: VX-150 vs Placebo; Test type: Superiority; p < 0.0001, Mixed-effects Model for Repeated Measure; Least Squares (LS) Mean Difference = -1.085, 95% CI 2-sided [-1.876 to -0.293]

2. Secondary Outcome: Percentage of Participants With Greater Than or Equal to (>=) 30 Percent (%) Reduction in the Weekly Average of Daily Pain Intensity on the 11-Point NRS
Description: Pain intensity was evaluated using the 11-point NRS (where 0 signified no pain and 10 signified worst imaginable pain) during the last 24 hours on the NRS each evening. Higher score indicates greater level of pain. Percentage of participants >= 30% reduction in the weekly average of daily pain intensity on the 11-Point NRS were reported.
Time Frame: From Baseline at Week 6
Population: FAS. Here, 'overall number of participants analyzed' signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | VX-150 | Placebo
Number analyzed (Participants) | 40 | 34
percentage of participants | 45.0 | 26.5

3. Secondary Outcome: Percentage of Participants With >=50% Reduction in the Weekly Average of Daily Pain Intensity on the 11-Point NRS
Description: Pain intensity was evaluated using the 11-point NRS (where 0 signified no pain and 10 signified worst imaginable pain) during the last 24 hours on the NRS each evening. Higher score indicates greater level of pain. Percentage of participants >= 50% reduction in the weekly average of daily pain intensity on the 11-Point NRS were reported.
Time Frame: From Baseline at Week 6
Population: FAS. Here, 'overall number of participants analyzed' signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | VX-150 | Placebo
Number analyzed (Participants) | 40 | 34
percentage of participants | 32.5 | 17.6

4. Secondary Outcome: Change in the Daily Sleep Interference Scale (DSIS)
Description: Pain-associated sleep interference was assessed using DSIS, based on an 11-point scale (where 0 signified none: pain does not interfere with sleep and 10 signified severe: pain completely interferes with sleep, unable to sleep). Higher score indicates greater pain associated sleep interference.
Time Frame: From Baseline at Week 6
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | VX-150 | Placebo
Number analyzed (Participants) | 46 | 43
units on a scale | -1.777 (0.276) | -0.665 (0.289)
Statistical Analysis 1: Comparison: VX-150 vs Placebo; Test type: Superiority; p < 0.0001, Mixed-effects Model for Repeated Measure; LS Mean Difference = -1.111, 95% CI 2-sided [-1.911 to -0.312]

5. Secondary Outcome: Percentage of Participants Categorized as Improved on the Patient Global Impression of Change (PGIC) Scale
Description: PGIC scale evaluated the change in activity limitations, symptoms, emotions, and overall quality of life (QoL) related to the participants painful condition on 7-point scale from 1 (improved) to 7 (worse). Participants were categorized as following: scale from 1 - 2 were categorized as "improved", scale from 3 - 4 as "no change" and scale from 5 - 7 were categorized as "worse". Percentage of participants categorized as improved on PGIC scale at week 6 were reported for this outcome measure.
Time Frame: At Week 6
Population: FAS. Here, 'overall number of participants analyzed' signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | VX-150 | Placebo
Number analyzed (Participants) | 43 | 37
percentage of participants | 39.5 | 13.5

6. Secondary Outcome: Change in Pain Intensity on the 11-Point NRS
Description: Pain intensity was evaluated using the 11-point NRS (where 0 signified no pain and 10 signified worst imaginable pain) during the last 24 hours on the NRS each evening. Higher score indicates greater level of pain. Higher score indicates greater level of pain.
Time Frame: From Baseline at Week 6
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | VX-150 | Placebo
Number analyzed (Participants) | 46 | 43
units on a scale | -1.7 (0.3) | -1.1 (0.3)
Statistical Analysis 1: Comparison: VX-150 vs Placebo; Test type: Superiority; p < 0.0001, Mixed-effects Model for Repeated Measure; LS Mean Difference = -0.6, 95% CI 2-sided [-1.5 to 0.3]

7. Secondary Outcome: Pre-dose Plasma Concentration (Ctrough) of VRT-1207355 and the Metabolite VRT-1268114
Time Frame: Pre-dose at Day 7
Population: Pharmacokinetic (PK) set included participants who received at least 1 dose of study drug and for whom the primary PK data was considered to be sufficient and interpretable.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | VX-150
Number analyzed (Participants) | 12
microgram per milliliter (mcg/mL)
  VRT-1207355 | 3.89 (2.73)
  VRT-1268114 | 1.35 (0.752)

8. Secondary Outcome: Number of Participants With Clinically Meaningful Findings in Columbia Suicide Severity Rating Scale (C-SSRS) Responses
Description: The C-SSRS is an interview-based rating scale was evaluated through a series of questions about suicidal thoughts and behaviors with the possible answers yes or no. Yes represents a worse outcome. Clinically Meaningfulness of C-SSRS responses were judged by investigator based on answers received from participants.
Time Frame: Day 1 up to Week 10
Population: Safety Set included all participants who have received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | VX-150 | Placebo
Number analyzed (Participants) | 46 | 43
participants | 0 | 0

9. Secondary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 10
Population: Safety set included all participants who had received at least 1 dose of the study drug.
Measure: Number; unit: participants
Arm/Group | VX-150 | Placebo
Number analyzed (Participants) | 46 | 43
participants
  Participants with AEs | 29 | 24
  Participants with SAEs | 0 | 3

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 10
Arm/Group | VX-150 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/46 | 3/43
Other Adverse Events (participants affected / at risk) | 16/46 | 7/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VX-150 (N=46) | Placebo (N=43)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VX-150 (N=46) | Placebo (N=43)
Dry mouth (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0
Headache (Nervous system disorders) | 11 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/22/NCT03304522/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT03304522/SAP_001.pdf